CLINICAL TRIAL: NCT04033042
Title: Performance and Safety Evaluation of a Novel Non-invasive Glucose Monitoring Device and Evaluation of the Instructions for Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RSP Systems A/S (Industry)
Collaborators: Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: RSP-21
Record Dates: First submitted 2019-07-15; First posted 2019-07-25 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus
Keywords: Non-invasive glucose monitoring; Raman spectroscopy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Masking Description: One group will receive the instructions for use and the other will not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protocol 1 (Experimental): RSP-21 Subjects will perform daily measurements on the IMD (Prototype 0.5) in addition to capillary reference measurements for 41 days.
  Interventions: Device: Prototype 0.5
- Protocol 2 (Experimental): RSP-21 Subjects will perform daily measurements on the IMD (Prototype 0.5) in addition to capillary reference measurements for 41 days.
  One group of subjects will receive training in the use of the device the other will not. Both groups will receive the instructions for use.
  Interventions: Device: Prototype 0.5

INTERVENTIONS:
Device: Prototype 0.5 — Subjects will perform daily measurements on the IMD (Prototype 0.5) for 41 days.

SUMMARY:
The aim of the study is to demonstrate the safety and performance of a novel non-invasive glucose monitoring device, to collect data and reference measurements for establishment of calibration models and to evaluate the instructions for use for the device. This study will be an explorative study with 10 study subjects.

DETAILED DESCRIPTION:
The Investigational Medical Device (IMD) for this investigation is the Prototype 0.5 (P0.5) developed and manufactured by RSP Systems (RSP). The device is intended for non-invasive interstitial intermittent glucose monitoring in persons (age 18 and older) with diabetes. The technology relies on the well-established capacities of Raman spectroscopy for directly detecting glucose subcutaneously. The Raman spectroscopy physical principle relies on the fact that when laser light of a given wavelength interferes with a molecule, a small fraction of the incident light will interact with the vibrational states of the molecule, causing the photons to lose a portion of their energy which will change the wavelength of the light. The scattered light will be collected by the optical probe head and analyzed with advanced algorithms to correlate the signal to glucose concentrations. Data collected from the IMD will be paired with validated glucose reference values collected by the finger sticking method.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ≥18 years of age
* Individuals diagnosed with type 1 diabetes. Gestational diabetes excluded
* Skin phototype 1-4
* Willing to perform up to 12 finger sticks during each day of out-patient measurements and up to 40 finger sticks at the two in-clinic study days
* Wireless internet connection at home to be used in the study

Exclusion Criteria:

* For female subjects: Pregnancy or subject is attempting to conceive or not willing and able to practice NCA approved birth control during the study duration
* For female subjects: breastfeeding
* Subjects currently participating in another study
* Subjects not able to understand and read German
* In investigator's opinion, subject is not able to follow instructions provided and as specified in the protocol
* Subject not able to hold hand/arm steady (including tremors and Parkinson's Disease)
* Extensive skin changes, tattoos or diseases on right hand thenar (sensor application site)
* Known allergy to medical grade alcohol
* Hemodialysis
* Systemic or topical administration of glucocorticoids at the right hand for the past 7 days or during the study period expected
* Medical history or any condition that may, in the opinion of the investigator compromise the subject's ability to participate
* Comorbidity or concomitant medical condition which, in the opinion of the Investigator, could interfere with the study or present a risk to the safety or welfare of the subject or study staff
* Severe diabetes related complications such as advanced autonomic neuropathy, kidney disease, foot ulcers, legal blindness, or symptomatic cardiovascular disease as evidenced by a history of cardiovascular episode(s)
* Dependency from the sponsor or the clinical investigator (e.g. co-workers of the sponsor, the study site, and/ or their families)
* Severe hypoglycemia resulting in seizure or loss of consciousness in the 3 months prior to enrollment
* Hypoglycemia unawareness
* Subjects who have participated in the study IDT-1639-RO

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Measurement accuracy | 4 months
  Accuracy of measurements performed on the IMD will be evaluated by data from subjects. Data will be analyzed by Mean Absolute Relative Difference (MARD).
Risk/benefit analysis | 4 months
  Risk/benefit analysis based on reported Adverse Device Effects and Serious Adverse Device Effects and the clinical performance safety profile.

SECONDARY OUTCOMES:
Review of IFU based on clinical performance. | 4 months
  Adequacy of IFU will be evaluated based on differences in clinical performance in two groups with and without personal training.
Review of IFU based on number of safety events. | 4 months
  Adequacy of IFU will be evaluated based on differences in safety events in two groups with and without personal training.
Number of encountered Device Deficiencies | 4 months
  Evaluation of device function with respect to identity, quality, durability, reliability, safety and performance

CONTACTS AND LOCATIONS:
Overall Officials: Guido Freckman, Principal Investigator — IfDT
Locations (1):
- Institut für Diabetes-Technologie Forschungs- und Entwicklungs-gesellschaft mbH an der Universität Ulm (IDT), Ulm, Germany

IPD SHARING:
Plan to Share IPD: No